CLINICAL TRIAL: NCT02187159
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled Study of DS-5565 for Treatment of Pain Associated With Fibromyalgia
Brief Title: Treatment of Pain Associated With Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS5565-A-E311; 2013-005163-10 (EudraCT Number)
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Pain Associated With Fibromyalgia
Keywords: pain; fibromyalgia
MeSH Terms: conditions — Pain; Fibromyalgia | interventions — mirogabalin; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DS-5565 QD (Experimental): Participants take one each of placebo tablet and capsule in the morning, and one DS-5565 tablet once daily (QD) with a placebo capsule in the evening
  Interventions: Drug: DS-5565; Drug: Placebo tablet; Drug: Placebo capsule
- DS-5565 BID (Experimental): Participants take one DS-5565 tablet and one placebo capsule, twice daily (BID)
  Interventions: Drug: DS-5565; Drug: Placebo capsule
- Pregabalin (Active Comparator): Participants take one pregabalin capsule and one placebo tablet BID
  Interventions: Drug: Pregabalin; Drug: Placebo tablet
- Placebo (Placebo Comparator): Participants take one each of placebo tablet and capsule BID
  Interventions: Drug: Placebo tablet; Drug: Placebo capsule

INTERVENTIONS:
Drug: DS-5565 — DS-5565 15 mg tablet for oral administration
  Other Names: mirogabalin
  Arms: DS-5565 BID; DS-5565 QD
Drug: Pregabalin — Pregabalin 150 mg capsule for oral administration
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo tablet — Placebo tablet (matching DS5565) for oral administration
  Other Names: Placebo matching DS-5565
  Arms: DS-5565 QD; Placebo; Pregabalin
Drug: Placebo capsule — Placebo capsule (matching pregabalin) for oral administration
  Other Names: Placebo matching pregabalin
  Arms: DS-5565 BID; DS-5565 QD; Placebo

SUMMARY:
The main objective of this trial is to compare change in weekly average daily pain score (ADPS) from baseline to Week 13 in participants receiving either dose of DS-5565 versus placebo. Weekly ADPS is based on daily pain scores reported by the participant that best describes his or her worst pain over the previous 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to give written informed consent
* Able to complete subject-reported questionnaires per the investigator's judgment
* At screening, subjects must meet the 1990 American College of Rheumatology (ACR) criteria for FM, i.e. widespread pain present for at least 3 months and pain in at least 11 of 18 specific tender point sites. In addition, the 2010 ACR criteria must be met:
* Widespread pain index (WPI) ≥ 7 and symptom severity (SS) scale score ≥ 5, or WPI 3 to 6 and SS scale score ≥ 9
* Symptoms have been present at a similar level for at least 3 months
* The subject does not have a disorder that would otherwise explain the pain
* ADPS of ≥ 4 on the 11-point numeric rating scale (NRS) over the past 7 days prior to randomization (based on completion of at least 4 daily pain diaries during the 7-day baseline period prior to randomization)
* Subject must have documented evidence of a fundoscopic examination (with pupil dilation) within 12 months prior to screening or at screening.
* Women of child-bearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy during the study and for 4 weeks after study completion.

Exclusion Criteria:

* Clinically significant unstable neurologic, psychiatric, ophthalmologic, hepatobiliary, respiratory, or hematologic illness or unstable cardiovascular disease (e.g. severe hypotension, uncontrolled cardiac arrhythmia, or myocardial infarction) or any other concurrent disease within 12 months prior to screening that in the opinion of the investigator would interfere with study participation or assessment of safety and tolerability
* Anticipation of initiation or significant change to normal daily exercise routines or need for ongoing use of concomitant medications or non-pharmacological pain management techniques that may confound assessments of efficacy and/or safety
* Unable to undergo pre-study washout of prohibited concomitant medications
* Subjects who are at risk of suicide as defined by their responses to the Columbia-Suicide Severity Rating Scale (C-SSRS) or in the opinion of the investigator. Note: Patients answering "yes" to any of the questions about active suicidal ideation/intent/behaviors occurring within the past 12 months must be excluded (C-SSRS Suicide Ideation section - Questions 3, 4, or 5; C-SSRS Suicidal Behavior section, any of the suicide behaviors questions). Such patients should be referred immediately to a mental health professional for appropriate evaluation.
* Current severe or uncontrolled major depressive disorder or anxiety disorders as assessed by the Mini-international Neuropsychiatric Interview (MINI) mild to moderate major depression or anxiety disorders are permitted provided that the investigator assesses the patient as clinically stable and appropriate for entry into the study.
* Any diagnosis of lifetime bipolar disorder or psychotic disorder
* Subjects with pain due to other conditions (e.g. diabetic peripheral neuropathic pain or post-herpetic neuralgia) that in the opinion of the investigator, would confound assessment or self-evaluation of the pain associated with FM.
* Subjects with pain due to any widespread inflammatory musculoskeletal disorder (e.g. rheumatoid arthritis, lupus) or widespread rheumatic disease other than FM.
* Abuse or dependence of prescription medications, street drugs, or alcohol within the last 1 year
* Any history of a malignancy other than basal cell carcinoma within the past 5 years
* A diagnosis of untreated sleep apnea or initiation of treatment for sleep apnea within the past 3 months
* Pregnancy or breast-feeding, or intent to become pregnant during the study period
* Subject is currently enrolled in or has not yet completed at least 30 days since ending another investigational device or drug study or is receiving other investigational agents.
* Known hypersensitivity to alpha2-delta (α2δ) ligands or other components of the study medications. Note: Prior exposure to DS-5565 is allowed, as long as hypersensitivity to DS-5565 was not observed.
* Subjects who are unlikely to comply with the protocol (e.g. uncooperative attitude, inability to return for subsequent visits) and/or otherwise considered by the investigator to be unlikely to complete the study.
* Abnormal investigative tests (i.e. electrocardiograms [ECGs]) and laboratory values judged by the investigator to be clinically significant at screening, with particular focus on: a. Abnormal renal function defined as calculated creatinine clearance (CrCl) < 60 mL/min determined by the central laboratory using the modified Cockcroft-Gault equation; blood urea nitrogen> 1.5 × upper limit of normal (ULN); creatine kinase > 3.0 × ULN; serum creatinine > 1.6 mg/dL (> 141.4 μmol/L); b. Abnormal liver function defined as aspartate aminotransferase (AST) > 2.0 × ULN, alanine aminotransferase (ALT) > 2.0 × ULN; alkaline phosphatase > 1.5 × ULN; total bilirubin> 1.2 × ULN. If a subject has total bilirubin > 1.2 ULN, unconjugated and conjugated bilirubin fractions should be analyzed and only subjects documented to have Gilbert's syndrome may be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1270 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-07-07 (Actual); Study Completion 2016-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (174):
- United States (84):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Fresno, California
  - Glendale, California
  - Orange, California
  - Oxnard, California
  - Richmond, California
  - Sacramento, California
  - San Diego, California
  - Santa Ana, California
  - Santa Barbara, California
  - Simi Valley, California
  - New London, Connecticut
  - Bradenton, Florida
  - Brandon, Florida
  - DeBary, Florida
  - Fort Myers, Florida
  - Hialeah, Florida
  - Homestead, Florida
  - Lake Mary, Florida
  - Miami, Florida
  - North Miami, Florida
  - Ocala, Florida
  - Plant City, Florida
  - Tampa, Florida
  - Alpharetta, Georgia
  - Atlanta, Georgia
  - Columbus, Georgia
  - Savannah, Georgia
  - Boise, Idaho
  - Meridian, Idaho
  - Chicago, Illinois
  - Gurnee, Illinois
  - Naperville, Illinois
  - Evansville, Indiana
  - West Des Moines, Iowa
  - Shawnee Mission, Kansas
  - Wichita, Kansas
  - Lexington, Kentucky
  - Monroe, Louisiana
  - Traverse City, Michigan
  - Jackson, Mississippi
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Brooklyn, New York
  - Manhasset, New York
  - New York, New York
  - Staten Island, New York
  - Benson, North Carolina
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Garfield Heights, Ohio
  - Middleburg Heights, Ohio
  - Tiffin, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Salem, Oregon
  - Duncansville, Pennsylvania
  - Warwick, Rhode Island
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Greer, South Carolina
  - Rock Hill, South Carolina
  - Bristol, Tennessee
  - Knoxville, Tennessee
  - New Tazewell, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Sealy, Texas
  - Sugar Land, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Kirkland, Washington
  - Charleston, West Virginia
- Australia (11):
  - Camperdown, New South Wales
  - Campsie, New South Wales
  - Coffs Harbour, New South Wales
  - St Leonards, New South Wales
  - Maroochydore, Queensland
  - Sherwood, Queensland
  - Southport, Queensland
  - Woodsville, South Australia
  - Hobart, Tasmania
  - Clayton, Victoria
  - Malvern East, Victoria
- Bulgaria (8):
  - Burgas
  - Pleven
  - Plovdiv
  - Rousse
  - Sevlievo
  - Sofia
  - Targovishte
  - Varna
- Estonia (2):
  - Tallinn
  - Tartu
- Hungary (8):
  - Balassagyarmat
  - Budapest
  - Debrecen
  - Esztergom
  - Kistarcsa
  - Nyíregyháza
  - Szeged
  - Veszprém
- India (7):
  - Ahmedabad, Gujarat
  - Surat, Gujarat
  - Bangalore, Karnataka
  - Hubli, Karnataka
  - Pune, Maharashtra
  - Jaipur, Rajasthan
  - Lucknow, VP
- Latvia (7):
  - Baldone
  - Balvi
  - Jēkabpils
  - Liepāja
  - Ogre
  - Riga
  - Ventspils
- New Zealand (5):
  - Auckland
  - Hamilton
  - Nelson
  - Tauranga
  - Wellington
- Romania (5):
  - Bacau
  - Bucharest
  - Cluj-Napoca
  - Oradea
  - Târgu Mureş
- Russia (10):
  - Ivanovo
  - Krasnoyarsk
  - Moscow
  - Nizhny Novgorod
  - Orenburgsky
  - Pyatigorski
  - Saint Petersburg
  - Stavropol
  - Vladikavkaz
  - Yaroslav
- Slovakia (7):
  - Banská Bystrica
  - Bratislava
  - Dubnica nad Váhom
  - Galanta
  - Krompachy
  - Piešťany
  - Prešov
- United Kingdom (20):
  - Reading, Berkshire
  - Penzance, Cornwall
  - Chesterfield, Derbyshire
  - Poole, Dorset
  - Romford, Essex
  - Blackpool, Lancashire
  - Thornton-Cleveleys, Lancashire
  - Wigan, Lancashire
  - Salford, Manchester
  - Southport, Merseyside
  - Wellingborough, Northamptonshire
  - Barnsley, South Yorkshire
  - Cannock, Staffordshire
  - North Shields, TYNE and WEAR
  - Atherstone, Warwickshire
  - Dudley, WEST Midlands
  - Belfast
  - Leeds
  - Manchester
  - Torpoint

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Arnold LM, Whitaker S, Hsu C, Jacobs D, Merante D. Efficacy and safety of mirogabalin for the treatment of fibromyalgia: results from three 13-week randomized, double-blind, placebo- and active-controlled, parallel-group studies and a 52-week open-label extension study. Curr Med Res Opin. 2019 Oct;35(10):1825-1835. doi: 10.1080/03007995.2019.1629757. Epub 2019 Jul 9. PMID 31284771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2280 participants who met all inclusion criteria and no exclusion criteria were enrolled from 19 Nov 2014 to 07 July 2016 at 178 sites. Of the 2280 participants enrolled, 1270 participants were randomized.
Pre-assignment Details: Eligible participants were randomized in a 1:1:1:1 ratio to either DS5565 15 mg QD, DS5565 15 mg BID, placebo, or pregabalin 150 mg BID.
Groups:
- Placebo: Participants who received oral pregabalin placebo and DS5565 placebo twice daily (BID).
- Pregabalin 150 mg BID: Participants who received oral pregabalin 150 mg twice daily (BID).
- DS-5565 15 mg QD: Participants who received oral DS5565 15 mg once daily (QD).
- DS-5565 15 mg BID: Participants who received DS-5565 15 mg twice daily (BID).
Period: Overall Study
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Started | 318 | 317 | 318 | 317
Completed | 249 | 238 | 241 | 221
Not Completed | 69 | 79 | 77 | 96
Not completed — Protocol Violation | 4 | 6 | 3 | 4
Not completed — Lack of Efficacy | 10 | 5 | 4 | 7
Not completed — Adverse Event | 28 | 33 | 42 | 50
Not completed — Withdrawal by Subject | 24 | 28 | 25 | 26
Not completed — Other | 3 | 7 | 3 | 9

BASELINE CHARACTERISTICS:
Population: Demographics at baseline were assessed in the Randomized Analysis Set.
Groups:
- Placebo: Participants take one each of placebo tablet and capsule BID)
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin | DS-5565 QD | DS-5565 BID | Total
Number analyzed (Participants) | 318 | 317 | 318 | 317 | 1270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 289 | 287 | 286 | 284 | 1146
  >=65 years | 29 | 30 | 32 | 33 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (11.43) | 50.9 (11.58) | 50.2 (11.85) | 50.6 (11.46) | 50.5 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 290 | 288 | 295 | 287 | 1160
  Male | 28 | 29 | 23 | 30 | 110
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 7 | 8 | 8 | 10 | 33
  Latvia | 7 | 9 | 6 | 10 | 32
  Romania | 9 | 11 | 6 | 5 | 31
  Hungary | 5 | 7 | 6 | 7 | 25
  United States | 188 | 188 | 188 | 188 | 752
  United Kingdom | 39 | 38 | 38 | 38 | 153
  Slovakia | 14 | 7 | 9 | 11 | 41
  Australia | 5 | 5 | 5 | 5 | 20
  Bulgaria | 16 | 19 | 22 | 17 | 74
  Estonia | 6 | 5 | 6 | 4 | 21
  India | 12 | 11 | 12 | 9 | 44
  Russia | 7 | 8 | 12 | 12 | 39
  Lithuania | 3 | 1 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 13 in Average Daily Pain Score (ADPS) in Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The patient reported pain intensity daily (over the past 24 hours) on a scale of 0 = no pain to 10 = worst possible pain. The daily pain scores were averaged over 7 days to calculate the weekly ADPS.
Time Frame: Baseline up to Week 13 postdose
Population: ADPS was assessed using the modified intent-to-treat (mITT) analysis set.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 315 | 311 | 315 | 313
units on a scale | -1.86 (0.130) | -2.47 (0.133) | -2.24 (0.133) | -2.09 (0.134)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg BID; Analysis was based on multiple imputation and pattern mixture model with delta shifting; Test type: Superiority; p = 0.0008, Difference of means; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-0.97 to -0.25], Standard Error of Mean 0.183
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg QD; Analysis was based on multiple imputation and pattern mixture model with delta shifting; Test type: Superiority; p = 0.0392, Difference of means; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.74 to -0.02], Standard Error of Mean 0.183
Statistical Analysis 3: Comparison: Placebo vs DS-5565 15 mg BID; Analysis was based on multiple imputation and pattern mixture model with delta shifting; Test type: Superiority; p = 0.2192, Difference of means; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.58 to 0.13], Standard Error of Mean 0.183
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Analysis was based on multiple imputation and pattern mixture model with delta shifting; Test type: Superiority; p = 0.2095, Difference of means; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.13 to 0.59], Standard Error of Mean 0.184
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Analysis was based on multiple imputation and pattern mixture model with delta shifting; Test type: Superiority; p = 0.0381, Difference of means; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [0.02 to 0.75], Standard Error of Mean 0.185

2. Secondary Outcome: Number of Participants Who Answered "Much Improved or Better" on the Patient Global Impression of Change (PGIC) Scale at Week 13 in Participants Receiving DS-5565, Pregabalin, or Placebo
Description: Patient-rated global impression of change (PGIC) on a categorical scale from 1 = very much improved to 7 = very much worse. The number of participants with "much improved or better" (≤2 scores) are reported.
Time Frame: Week 13 postdose
Population: PGIC was assessed using the modified intent-to-treat (mITT) analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 315 | 312 | 315 | 313
Participants | 91 | 141 | 116 | 117

3. Secondary Outcome: Change From Baseline to Week 13 in Fibromyalgia Index Questionnaire (FIQ) Total Score in Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The total FIQ score is composed of 10 items, with a maximum possible score of 100. The first item contains 11 questions related to physical functioning and are rated on a 4-point Likert-type scale, where 0 indicates 'always' and 3 indicates 'never'. The overall impact items are rated on a 0-7 scale for the number of days that the patient felt well and the number of days they were unable to work (including housework) because of fibromyalgia symptoms. The symptoms items are rated on visual analog scales (0-10 cm), with higher numbers indicated greater symptomatology. Final scores range from 0 (no impairment) to 10 (maximum impairment), where higher scores indicate worse outcome.
  For this outcome, the change in total FIQ score from baseline is being reported. Negative values indicate improvement from baseline in impairment.
Time Frame: Baseline up to Week 13 postdose
Population: FIQ was assessed using the modified intent-to-treat (mITT) analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 313 | 312 | 312 | 312
units on a scale | -13.88 (1.20) | -21.46 (1.22) | -17.41 (1.22) | -16.45 (1.24)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg BID; Analysis was based on multiple imputation and pattern mixture model with delta shifting; Test type: Superiority; p < 0.0001, Difference of means; Mean Difference (Final Values) = -7.67, 95% CI 2-sided [-10.71 to -4.44], Standard Error of Mean 1.598
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg QD; Analysis was based on multiple imputation and pattern mixture model with delta shifting; Test type: Superiority; p = 0.0289, Difference of means; Mean Difference (Final Values) = -3.52, 95% CI 2-sided [-6.68 to -0.36], Standard Error of Mean 1.613
Statistical Analysis 3: Comparison: Placebo vs DS-5565 15 mg BID; Analysis was based on multiple imputation and pattern mixture model with delta shifting; Test type: Superiority; p = 0.1148, Difference of means; Mean Difference (Final Values) = -2.56, 95% CI 2-sided [-5.75 to 0.62], Standard Error of Mean 1.625
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Analysis was based on multiple imputation and pattern mixture model with delta shifting; Test type: Superiority; p = 0.0125, Difference of means; Mean Difference (Final Values) = 4.05, 95% CI 2-sided [0.87 to 7.23], Standard Error of Mean 1.621
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Analysis was based on multiple imputation and pattern mixture model with delta shifting; Test type: Superiority; p = 0.0023, Difference of means; Mean Difference (Final Values) = 5.01, 95% CI 2-sided [1.78 to 8.24], Standard Error of Mean 1.647

4. Secondary Outcome: Number of Responders at Week 13 Among Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The number of participants with at least a 30% or 50% reduction in average daily pain score (ADPS) at Week 13 is reported.
Time Frame: Week 13 postdose
Population: Responder rates were assessed using the modified intent-to-treat (mITT) analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 315 | 312 | 315 | 313
Participants
  30% Responders | 113 | 139 | 123 | 118
  50% Responders | 61 | 90 | 79 | 68

5. Secondary Outcome: Change From Baseline to Week 13 in Multidimensional Fatigue Inventory (MFI-20) General Fatigue Score in Participants Receiving DS-5565, Pregabalin, or Placebo
Description: MFI is a validated 20-item, self-reported instrument designed to measure fatigue in the following dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. The respondent is asked to mark an 'X' in 1 of 5 boxes arranged linearly where 1 is 'Yes, that is true' and 5 is 'No, that is not true.' Each subscale consists of 4 items, 2 indicative for fatigue and 2 contraindicative. For the indicative questions, a high score indicates a high fatigue level and low scores indicate a low fatigue levels. Conversely, for the contraindicative questions a high score indicates a low fatigue level and a low score indicates a high fatigue level. Overall, respondents are rated on a scale of 0 (no fatigue) to 7 (high fatigue).
  For this outcome, the change from baseline in MFI-20 general fatigue subscale score is being reported. Negative values indicate an improvement in fatigue.
Time Frame: Baseline up to Week 13 postdose
Population: Multidimensional Fatigue Inventory (MFI-20) was assessed in the modified intent-to-treat (mITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 293 | 294 | 295 | 291
units on a scale | -1.4 (3.45) | -2.8 (3.99) | -2.3 (3.57) | -2.1 (3.45)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Difference in least squares means = -1.2, 95% CI 2-sided [-1.8 to -0.7], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0247, ANCOVA; Difference in least squares means = -0.6, 95% CI 2-sided [-1.2 to -0.1], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0411, ANCOVA; Difference in least squares means = -0.6, 95% CI 2-sided [-1.1 to -0.0], Standard Error of Mean 0.29
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0352, ANCOVA; Difference in least squares means = 0.6, 95% CI 2-sided [0.0 to 1.2], Standard Error of Mean 0.29
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0214, ANCOVA; Difference in least squares means = 0.7, 95% CI 2-sided [0.1 to 1.2], Standard Error of Mean 0.29

6. Secondary Outcome: Change From Baseline to Week 13 in Hospital Anxiety and Depression Scale (HADS) in Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The HADS questionnaire is a reliable, widely-used self-assessment scale to assess symptoms of anxiety and depression. The instrument consists of 7 questions related to anxiety and 7 related to depression, each rated on a 4-point scale (score of 0 to 3). Scores for anxiety and depression are independently summed to compute HADS-Anxiety and HADS-Depression subscale scores, with ranges from 0 (no anxiety/depression) to 21 (most severe anxiety/depression).
Time Frame: Baseline up to Week 13 postdose
Population: HADS was assessed using the modified intent-to-treat (mITT) analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 315 | 312 | 315 | 313
units on a scale
  Change from baseline to Week 13: Anxiety: number analyzed (Participants) | 293 | 294 | 295 | 291
  Change from baseline to Week 13: Anxiety | -0.5 (3.43) | -1.4 (3.47) | -0.7 (3.30) | -0.8 (3.31)
  Change from baseline to Week 13: Depression: number analyzed (Participants) | 293 | 294 | 295 | 291
  Change from baseline to Week 13: Depression | -0.8 (3.66) | -1.6 (3.86) | -1.1 (3.78) | -0.8 (3.83)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg BID; Anxiety: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0003, ANCOVA; Difference of least squares means = -0.9, 95% CI 2-sided [-1.5 to -0.4], Standard Error of Mean 0.26
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg QD; Anxiety: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.5066, ANCOVA; Difference of least squares means = -0.2, 95% CI 2-sided [-0.7 to 0.3], Standard Error of Mean 0.26
Statistical Analysis 3: Comparison: Placebo vs DS-5565 15 mg BID; Anxiety: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.1462, ANCOVA; Difference of least squares means = -0.4, 95% CI 2-sided [-0.9 to 0.1], Standard Error of Mean 0.26
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Anxiety: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0035, ANCOVA; Difference of least squares means = 0.8, 95% CI 2-sided [0.3 to 1.3], Standard Error of Mean 0.26
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Anxiety: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0338, ANCOVA; Difference in least squares means = 0.6, 95% CI 2-sided [0.0 to 1.1], Standard Error of Mean 0.26
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 150 mg BID; Depression: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0116, ANCOVA; Difference in least squares means = -0.7, 95% CI 2-sided [-1.3 to -0.2], Standard Error of Mean 0.28
Statistical Analysis 7: Comparison: Placebo vs DS-5565 15 mg QD; Depression: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.7085, ANCOVA; Difference of least squares means = -0.1, 95% CI 2-sided [-0.7 to 0.4], Standard Error of Mean 0.28
Statistical Analysis 8: Comparison: Placebo vs DS-5565 15 mg BID; Depression: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.9392, ANCOVA; Difference in least squares means = 0.0, 95% CI 2-sided [-0.5 to 0.6], Standard Error of Mean 0.28
Statistical Analysis 9: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Depression: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0311, ANCOVA; Difference in least squares means = 0.6, 95% CI 2-sided [0.1 to 1.2], Standard Error of Mean 0.28
Statistical Analysis 10: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Depression: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0094, ANCOVA; Difference in least squares means = 0.7, 95% CI 2-sided [0.2 to 1.3], Standard Error of Mean 0.28

7. Secondary Outcome: Change From Baseline to Week 13 in Short Form 36 (SF-36) in Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The SF-36 is a 36-question health survey that measures functional health and well-being from the participant's point of view. It is a measure of physical and mental health used across various disease areas, including fibromyalgia. The SF-36 scale ranges from 0 to 100 where lower scores indicate more disability (worse health) and higher scores represent less disability (better health). The physical component summary (PCS) and mental component summary (MCS) scores are reported.
Time Frame: Baseline up to Week 13 postdose
Population: This outcome was assessed using the modified intent-to-treat analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 315 | 312 | 315 | 313
units on a scale
  Change from baseline to Week 13:Physical Component: number analyzed (Participants) | 293 | 293 | 295 | 291
  Change from baseline to Week 13:Physical Component | 4.395 (6.81) | 5.815 (8.03) | 5.000 (7.76) | 4.833 (7.18)
  Change from baseline to Week 13: Mental Component: number analyzed (Participants) | 293 | 293 | 295 | 291
  Change from baseline to Week 13: Mental Component | 1.371 (9.43) | 3.093 (8.93) | 1.675 (9.94) | 1.198 (8.37)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg BID; Physical Component: Placebo vs Pregabalin; Test type: Superiority; p = 0.0373, ANCOVA; Difference in least squares means = 1.256, 95% CI 2-sided [0.074 to 2.439], Standard Error of Mean 0.6027
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg QD; Physical Component: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.5458, ANCOVA; Difference of least squares means = 0.364, 95% CI 2-sided [-0.817 to 1.545], Standard Error of Mean 0.6020
Statistical Analysis 3: Comparison: Placebo vs DS-5565 15 mg BID; Physical Component: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.6968, ANCOVA; Difference in least squares means = 0.235, 95% CI 2-sided [-0.949 to 1.420], Standard Error of Mean 0.6038
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Physical Component: Pregabalin vs DS-5565 15 mg QD; Test type: Superiority; p = 0.1379, ANCOVA; Difference in least squares means = -0.893, 95% CI 2-sided [-2.073 to 0.287], Standard Error of Mean 0.6014
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Physical Component: Pregabalin vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0908, ANCOVA; Difference in least squares means = -1.021, 95% CI 2-sided [-2.205 to 0.163], Standard Error of Mean 0.6033
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 150 mg BID; Mental Component: Placebo vs Pregabalin; Test type: Superiority; p = 0.0068, ANCOVA; Difference in least squares means = 1.890, 95% CI 2-sided [0.523 to 3.256], Standard Error of Mean 0.6965
Statistical Analysis 7: Comparison: Placebo vs DS-5565 15 mg QD; Mental Component: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.5594, ANCOVA; Difference in least squares means = 0.406, 95% CI 2-sided [-0.959 to 1.771], Standard Error of Mean 0.6956
Statistical Analysis 8: Comparison: Placebo vs DS-5565 15 mg BID; Mental Component: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.9736, ANCOVA; Difference in least squares means = 0.023, 95% CI 2-sided [-1.346 to 1.392], Standard Error of Mean 0.6979
Statistical Analysis 9: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Mental Component: Pregabalin vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0331, ANCOVA; Difference in least squares means = -1.484, 95% CI 2-sided [-2.848 to -0.119], Standard Error of Mean 0.6953
Statistical Analysis 10: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Mental Component: Pregabalin vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0076, ANCOVA; Difference in least squares means = -1.867, 95% CI 2-sided [-3.235 to -0.498], Standard Error of Mean 0.6976

8. Secondary Outcome: Change From Baseline to Week 13 in EuroQol Five Dimensions Questionnaire (EQ-5D) in Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The EQ-5D is an instrument that shows high construct validity and responsiveness in patients with chronic pain and has been used specifically in fibromyalgia. The EQ-5D includes a descriptive section with 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each with a scale that ranges from 0 (no problems) to 5 (extreme problems). These 5 dimensions are combined into an overall health utilities index, and a numeric rating scale (100 mm visual analog scale) that measures perception of overall health, with 0 indicating worst health and 100 representing best imaginable health. A summary index with a maximum total score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum total score of 1 indicates the best health outcome.
  For this outcome, the change from baseline in total EQ-5D score is being reported. Positive values indicate an improvement in health.
Time Frame: Baseline up to Week 13 postdose
Population: The EQ-5D was assessed using the modified intent-to-treat (mITT) analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 293 | 292 | 295 | 291
units on a scale | 0.060 (0.18) | 0.10 (0.19) | 0.08 (0.17) | 0.07 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0201, ANCOVA; Difference in least squares means = 0.0309, 95% CI 2-sided [0.0048 to 0.0570], Standard Error of Mean 0.01328
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.1798, ANCOVA; Difference of least squares means = 0.0178, 95% CI 2-sided [-0.0082 to 0.0438], Standard Error of Mean 0.01324
Statistical Analysis 3: Comparison: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.5922, ANCOVA; Difference of least squares means = 0.0071, 95% CI 2-sided [-0.0189 to 0.0332], Standard Error of Mean 0.01329
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.3221, ANCOVA; Difference in least squares means = -0.0131, 95% CI 2-sided [-0.0392 to 0.0129], Standard Error of Mean 0.01326
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0739, ANCOVA; Difference in least squares means = -0.0238, 95% CI 2-sided [-0.0499 to 0.0023], Standard Error of Mean 0.01330

9. Secondary Outcome: Change From Baseline to Week 13 in Average Daily Sleep Interference Score (ADSIS) in Participants Receiving DS-5565, Pregabalin, or Placebo
Description: Pain-associated sleep interference was assessed using electronic daily diaries using an 11-point numeric rating scale (NRS) for pain, ranging from 0 (pain does not interfere with sleep) to 10 (pain completely interferes with sleep, unable to sleep). ADSIS is the mean value of all available recordings of the respective week.
Time Frame: Baseline up to Week 13 postdose
Population: Pain-associated sleep interference was assessed using the modified intent-to-treat (mITT) analysis set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 315 | 312 | 315 | 313
units on a scale | -1.92 (0.11) | -2.41 (0.11) | -2.48 (0.11) | -2.44 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0015, Mixed Models Analysis; Difference in least squares means = -0.49, 95% CI 2-sided [-0.79 to -0.19], Standard Error of Mean 0.153
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Difference in least squares means = -0.56, 95% CI 2-sided [-0.86 to -0.26], Standard Error of Mean 0.153
Statistical Analysis 3: Comparison: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0008, Mixed Models Analysis; Difference in least squares means = -0.51, 95% CI 2-sided [-0.81 to -0.21], Standard Error of Mean 0.153
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.6464, Mixed Models Analysis; Difference in least squares means = -0.07, 95% CI 2-sided [-0.37 to 0.23], Standard Error of Mean 0.154
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.8543, Mixed Models Analysis; Difference in least squares means = -0.03, 95% CI 2-sided [-0.33 to 0.27], Standard Error of Mean 0.154

10. Secondary Outcome: The Number of Participants Reporting Optimal Sleep at Week 13 on the Medical Outcomes Study (MOS) Sleep Scale in Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The MOS sleep scale is a 12-item questionnaire from which the following subscales were derived: sleep disturbance (4 items), quantity of sleep/optimal sleep (1 item), snoring (1 item), awakening due to shortness of breath or due to headache (1 item), sleep adequacy (2 items), and somnolence (3 items). In addition, values for sleep disturbances index (9 items), optimal sleep scale (1 item), sleep quantity scale (1 item) were determine. Most subscales range from 0 to 100, where higher scores indicate more of the concept being measured (eg., higher sleep disturbance scores indicate greater sleep disturbances).
Time Frame: Week 13 postdose
Population: The MOS sleep scale outcome was assessed in the modified intent-to-treat (mITT) analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 315 | 312 | 315 | 313
Participants | 90 | 94 | 101 | 106

11. Secondary Outcome: Change From Baseline to Week 13 in the Brief Pain Inventory Short Form (BPI-SF) in Participants Receiving DS-5565, Pregabalin, or Placebo
Description: The BPI-SF measures pain severity and interference within the past 24 hours. Items are rated on an 11-point NRS from 0 to 10, where 0 indicates does not interfere and 10 indicates completely interferes. Severity score is the average of the responses to the 4 pain intensity items that assess the Worst/Least/Average pain in the last 24 hours and the Pain Right Now. The individual items being reported (using the same scale as noted above) are Severity, General Activity, Mood, Walking Ability, Normal Work, Relations With Other People, Sleep, and Enjoyment of Life. Percentage relief of treatment pain scale ranges from 100% (complete pain relief) to 0% (no pain relief) and higher percentages indicate better outcome. Interference % is the average of responses for General activity, Mood, Walking ability, Normal work, Relations with other people, Sleep, Enjoyment of life where 0% (no interference) to 100% (completely interferes) and negative (ie. lower) percentages indicate better outcomes.
Time Frame: Baseline up to Week 13 postdose
Population: BFI-SF was assessed using the modified intent-to-treat (mITT) analysis set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 315 | 312 | 315 | 313
units on a scale
  Worst pain: number analyzed (Participants) | 244 | 234 | 236 | 220
  Worst pain | -1.7 (2.36) | -2.6 (2.37) | -2.2 (2.55) | -2.1 (2.30)
  Least pain: number analyzed (Participants) | 244 | 234 | 236 | 220
  Least pain | -1.4 (2.53) | -1.9 (2.37) | -1.5 (2.53) | -1.6 (2.25)
  Average pain: number analyzed (Participants) | 244 | 234 | 236 | 220
  Average pain | -1.5 (2.13) | -2.1 (2.15) | -1.8 (2.15) | -1.8 (1.96)
  Pain right now: number analyzed (Participants) | 244 | 234 | 236 | 220
  Pain right now | -1.8 (2.76) | -2.8 (2.48) | -2.3 (2.54) | -2.2 (2.40)
  Severity score: number analyzed (Participants) | 244 | 234 | 236 | 220
  Severity score | -1.59 (2.17) | -2.33 (2.08) | -1.96 (2.17) | -1.91 (1.95)
  Relief (%) by treatment of pain: number analyzed (Participants) | 244 | 234 | 236 | 220
  Relief (%) by treatment of pain | 20.1 (33.69) | 31.1 (33.15) | 24.2 (33.26) | 25.9 (35.09)
  Interference (%): number analyzed (Participants) | 244 | 234 | 236 | 220
  Interference (%) | -14.79 (22.33) | -23.76 (21.81) | -19.97 (23.37) | -18.35 (20.68)
  General activity: number analyzed (Participants) | 244 | 234 | 236 | 220
  General activity | -1.6 (2.77) | -2.5 (2.63) | -2.1 (2.66) | -2.1 (2.53)
  Mood: number analyzed (Participants) | 244 | 234 | 236 | 220
  Mood | -1.3 (2.84) | -2.2 (2.65) | -1.6 (2.94) | -1.6 (2.65)
  Walking ability: number analyzed (Participants) | 244 | 234 | 236 | 220
  Walking ability | -1.5 (2.60) | -2.1 (2.79) | -1.8 (2.88) | -1.4 (2.60)
  Normal work: number analyzed (Participants) | 244 | 234 | 236 | 220
  Normal work | -1.6 (2.65) | -2.3 (2.70) | -1.9 (2.77) | -1.9 (2.60)
  Relations with other people: number analyzed (Participants) | 244 | 234 | 236 | 220
  Relations with other people | -1.2 (2.92) | -1.8 (2.92) | -1.6 (3.12) | -1.2 (2.85)
  Sleep: number analyzed (Participants) | 244 | 234 | 236 | 220
  Sleep | -1.9 (2.99) | -3.3 (2.83) | -3.1 (3.14) | -3.0 (2.80)
  Enjoyment of life: number analyzed (Participants) | 244 | 234 | 236 | 220
  Enjoyment of life | -1.3 (3.00) | -2.4 (2.85) | -1.9 (3.22) | -1.7 (2.98)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg BID; Worst pain: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0014, ANCOVA; Difference in least squares means = -0.6, 95% CI 2-sided [-1.0 to 0.2], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg QD; Worst pain: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.1285, ANCOVA; Difference of least squares means = -0.3, 95% CI 2-sided [-0.7 to 0.1], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: Placebo vs DS-5565 15 mg BID; Worst pain: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.6595, ANCOVA; Difference in least squares means = -0.1, 95% CI 2-sided [-0.5 to 0.3], Standard Error of Mean 0.19
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Worst pain: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0938, ANCOVA; Difference in least squares means = 0.3, 95% CI 2-sided [-0.1 to 0.7], Standard Error of Mean 0.19
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Worst pain: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0061, ANCOVA; Difference in least squares means = 0.5, 95% CI 2-sided [0.1 to 0.9], Standard Error of Mean 0.19
Statistical Analysis 6: Comparison: Placebo vs Pregabalin 150 mg BID; Least pain: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0235, ANCOVA; Difference in least squares means = -0.4, 95% CI 2-sided [-0.8 to -0.1], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Placebo vs DS-5565 15 mg QD; Least pain: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.3652, ANCOVA; Difference in least squares means = -0.2, 95% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.18
Statistical Analysis 8: Comparison: Placebo vs DS-5565 15 mg BID; Least pain: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.6885, ANCOVA; Difference in least squares means = -0.1, 95% CI 2-sided [-0.4 to 0.3], Standard Error of Mean 0.18
Statistical Analysis 9: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Least pain: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.1726, ANCOVA; Difference in least squares means = 0.2, 95% CI 2-sided [-0.1 to 0.6], Standard Error of Mean 0.18
Statistical Analysis 10: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Least pain: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0627, ANCOVA; Difference in least squares means = 0.3, 95% CI 2-sided [-0.0 to 0.7], Standard Error of Mean 0.18
Statistical Analysis 11: Comparison: Placebo vs Pregabalin 150 mg BID; Average pain: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0026, ANCOVA; Difference in least squares means = -0.5, 95% CI 2-sided [-0.8 to -0.2], Standard Error of Mean 0.16
Statistical Analysis 12: Comparison: Placebo vs DS-5565 15 mg QD; Average pain: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.1362, ANCOVA; Difference in least squares means = -0.2, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.16
Statistical Analysis 13: Comparison: Placebo vs DS-5565 15 mg BID; Average pain: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.4344, ANCOVA; Difference in least squares means = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.16
Statistical Analysis 14: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Average pain: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.1264, ANCOVA; Difference in least squares means = 0.2, 95% CI 2-sided [-0.1 to 0.6], Standard Error of Mean 0.16
Statistical Analysis 15: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Average pain: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0260, ANCOVA; Difference in least squares means = 0.4, 95% CI 2-sided [0.0 to 0.7], Standard Error of Mean 0.16
Statistical Analysis 16: Comparison: Placebo vs Pregabalin 150 mg BID; Pain right now: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0002, ANCOVA; Difference in least squares means = -0.7, 95% CI 2-sided [-1.1 to -0.4], Standard Error of Mean 0.20
Statistical Analysis 17: Comparison: Placebo vs DS-5565 15 mg QD; Pain right now: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0597, ANCOVA; Difference in least squares means = -0.4, 95% CI 2-sided [-0.8 to 0.0], Standard Error of Mean 0.20
Statistical Analysis 18: Comparison: Placebo vs DS-5565 15 mg BID; Pain right now: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.1198, ANCOVA; Difference in least squares means = -0.3, 95% CI 2-sided [-0.7 to 0.1], Standard Error of Mean 0.20
Statistical Analysis 19: Comparison: Placebo vs Pregabalin 150 mg BID; Severity score: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0006, ANCOVA; Difference in least squares means = -0.563, 95% CI 2-sided [-0.885 to -0.240], Standard Error of Mean 0.1644
Statistical Analysis 20: Comparison: Placebo vs DS-5565 15 mg QD; Severity score: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.1118, ANCOVA; Difference in least squares means = -0.261, 95% CI 2-sided [-0.583 to 0.061], Standard Error of Mean 0.1640
Statistical Analysis 21: Comparison: Placebo vs DS-5565 15 mg BID; Severity score: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.3870, ANCOVA; Difference in least squares means = -0.142, 95% CI 2-sided [-0.465 to 0.180], Standard Error of Mean 0.1646
Statistical Analysis 22: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Severity score: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0633, ANCOVA; Difference in least squares means = 0.302, 95% CI 2-sided [-0.020 to 0.624], Standard Error of Mean 0.1642
Statistical Analysis 23: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Severity score: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0108, ANCOVA; Difference in least squares means = 0.420, 95% CI 2-sided [0.097 to 0.744], Standard Error of Mean 0.1647
Statistical Analysis 24: Comparison: Placebo vs Pregabalin 150 mg BID; Relief by treatment of pain: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0020, ANCOVA; Difference in least squares means = 7.5, 95% CI 2-sided [2.7 to 12.2], Standard Error of Mean 2.41
Statistical Analysis 25: Comparison: Placebo vs DS-5565 15 mg QD; Relief by treatment of pain: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.2188, ANCOVA; Difference in least squares means = 3.0, 95% CI 2-sided [-1.8 to 7.7], Standard Error of Mean 2.41
Statistical Analysis 26: Comparison: Placebo vs DS-5565 15 mg BID; Relief by treatment of pain: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0991, ANCOVA; Difference in least squares means = 4.0, 95% CI 2-sided [-0.8 to 8.7], Standard Error of Mean 2.41
Statistical Analysis 27: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Relief by treatment of pain: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0611, ANCOVA; Difference in least squares means = -4.5, 95% CI 2-sided [-9.2 to 0.2], Standard Error of Mean 2.41
Statistical Analysis 28: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Relief by treatment of pain: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.1489, ANCOVA; Difference in least squares means = -3.5, 95% CI 2-sided [-8.2 to 1.2], Standard Error of Mean 2.41
Statistical Analysis 29: Comparison: Placebo vs Pregabalin 150 mg BID; Interference: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0006, ANCOVA; Difference in least squares means = -6.04, 95% CI 2-sided [-9.47 to -2.60], Standard Error of Mean 1.751
Statistical Analysis 30: Comparison: Placebo vs DS-5565 15 mg QD; Interference: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0193, ANCOVA; Difference in least squares means = -4.09, 95% CI 2-sided [-7.52 to -0.67], Standard Error of Mean 1.747
Statistical Analysis 31: Comparison: Placebo vs DS-5565 15 mg BID; Interference: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.3506, ANCOVA; Difference in least squares means = -1.64, 95% CI 2-sided [-5.07 to 1.80], Standard Error of Mean 1.752
Statistical Analysis 32: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Interference: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.2660, ANCOVA; Difference in least squares means = 1.94, 95% CI 2-sided [-1.48 to 5.37], Standard Error of Mean 1.748
Statistical Analysis 33: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Interference: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0122, ANCOVA; Difference in least squares means = 4.40, 95% CI 2-sided [0.96 to 7.84], Standard Error of Mean 1.754
Statistical Analysis 34: Comparison: Placebo vs Pregabalin 150 mg BID; General activity: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0119, ANCOVA; Difference in least squares means = -0.5, 95% CI 2-sided [-0.9 to -0.1], Standard Error of Mean 0.20
Statistical Analysis 35: Comparison: Placebo vs DS-5565 15 mg QD; General activity: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0659, ANCOVA; Difference in least squares means = -0.4, 95% CI 2-sided [-0.8 to 0.0], Standard Error of Mean 0.20
Statistical Analysis 36: Comparison: Placebo vs DS-5565 15 mg BID; General activity: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.5104, ANCOVA; Difference in least squares means = -0.1, 95% CI 2-sided [-0.5 to 0.3], Standard Error of Mean 0.20
Statistical Analysis 37: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; General activity: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.4934, ANCOVA; Difference in least squares means = 0.1, 95% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.20
Statistical Analysis 38: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; General activity: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0634, ANCOVA; Difference in least squares means = 0.4, 95% CI 2-sided [-0.0 to 0.8], Standard Error of Mean 0.20
Statistical Analysis 39: Comparison: Placebo vs Pregabalin 150 mg BID; Mood: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0007, ANCOVA; Difference in least squares means = -0.7, 95% CI 2-sided [-1.1 to -0.3], Standard Error of Mean 0.21
Statistical Analysis 40: Comparison: Placebo vs DS-5565 15 mg QD; Mood: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0837, ANCOVA; Difference in least squares means = -0.4, 95% CI 2-sided [-0.8 to 0.0], Standard Error of Mean 0.21
Statistical Analysis 41: Comparison: Placebo vs DS-5565 15 mg BID; Mood: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.2379, ANCOVA; Difference in least squares means = -0.2, 95% CI 2-sided [-0.7 to 0.2], Standard Error of Mean 0.21
Statistical Analysis 42: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Mood: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0980, ANCOVA; Difference in least squares means = 0.3, 95% CI 2-sided [-0.1 to 0.8], Standard Error of Mean 0.21
Statistical Analysis 43: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Mood: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0283, ANCOVA; Difference in least squares means = 0.5, 95% CI 2-sided [0.0 to 0.9], Standard Error of Mean 0.21
Statistical Analysis 44: Comparison: Placebo vs Pregabalin 150 mg BID; Walking ability: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.2179, ANCOVA; Difference in least squares means = -0.3, 95% CI 2-sided [-0.7 to 0.2], Standard Error of Mean 0.21
Statistical Analysis 45: Comparison: Placebo vs DS-5565 15 mg QD; Walking ability: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.6683, ANCOVA; Difference in least squares means = -0.1, 95% CI 2-sided [-0.5 to 0.3], Standard Error of Mean 0.21
Statistical Analysis 46: Comparison: Placebo vs DS-5565 15 mg BID; Walking ability: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.2247, ANCOVA; Difference in least squares means = 0.3, 95% CI 2-sided [-0.2 to 0.7], Standard Error of Mean 0.21
Statistical Analysis 47: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Walking ability: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.4198, ANCOVA; Difference in least squares means = 0.2, 95% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.21
Statistical Analysis 48: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Walking ability: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0146, ANCOVA; Difference in least squares means = 0.5, 95% CI 2-sided [0.1 to 0.9], Standard Error of Mean 0.21
Statistical Analysis 49: Comparison: Placebo vs Pregabalin 150 mg BID; Normal work: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0662, ANCOVA; Difference in least squares means = -0.4, 95% CI 2-sided [-0.8 to 0.0], Standard Error of Mean 0.21
Statistical Analysis 50: Comparison: Placebo vs DS-5565 15 mg QD; Normal work: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.2282, ANCOVA; Difference in least squares means = -0.3, 95% CI 2-sided [-0.7 to 0.2], Standard Error of Mean 0.21
Statistical Analysis 51: Comparison: Placebo vs DS-5565 15 mg BID; Normal work: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.7336, ANCOVA; Difference in least squares means = -0.1, 95% CI 2-sided [-0.5 to 0.3], Standard Error of Mean 0.21
Statistical Analysis 52: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Normal work: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.5240, ANCOVA; Difference in least squares means = 0.1, 95% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.21
Statistical Analysis 53: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Normal work: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.1349, ANCOVA; Difference in least squares means = 0.3, 95% CI 2-sided [-0.1 to 0.7], Standard Error of Mean 0.21
Statistical Analysis 54: Comparison: Placebo vs Pregabalin 150 mg BID; Relations with other people: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0464, ANCOVA; Difference in least squares means = -0.4, 95% CI 2-sided [-0.8 to -0.0], Standard Error of Mean 0.21
Statistical Analysis 55: Comparison: Placebo vs DS-5565 15 mg QD; Relations with other people: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0975, ANCOVA; Difference in least squares means = -0.3, 95% CI 2-sided [-0.7 to 0.1], Standard Error of Mean 0.21
Statistical Analysis 56: Comparison: Placebo vs DS-5565 15 mg BID; Relations with other people: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.6088, ANCOVA; Difference in least squares means = 0.1, 95% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.21
Statistical Analysis 57: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Relations with other people: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.7341, ANCOVA; Difference in least squares means = 0.1, 95% CI 2-sided [-0.3 to 0.5], Standard Error of Mean 0.21
Statistical Analysis 58: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Relations with other people: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0125, ANCOVA; Difference in least squares means = 0.5, 95% CI 2-sided [0.1 to 0.9], Standard Error of Mean 0.21
Statistical Analysis 59: Comparison: Placebo vs Pregabalin 150 mg BID; Sleep: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p < 0.0001, ANCOVA; Difference in least squares means = -1.0, 95% CI 2-sided [-1.4 to -0.5], Standard Error of Mean 0.23
Statistical Analysis 60: Comparison: Placebo vs DS-5565 15 mg QD; Sleep: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0003, ANCOVA; Difference in least squares means = -0.8, 95% CI 2-sided [-1.3 to -0.4], Standard Error of Mean 0.23
Statistical Analysis 61: Comparison: Placebo vs DS-5565 15 mg BID; Sleep: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0040, ANCOVA; Difference in least squares means = -0.7, 95% CI 2-sided [-1.1 to -0.2], Standard Error of Mean 0.23
Statistical Analysis 62: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Sleep: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.5801, ANCOVA; Difference in least squares means = 0.1, 95% CI 2-sided [-0.3 to 0.6], Standard Error of Mean 0.23
Statistical Analysis 63: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Sleep: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.1869, ANCOVA; Difference in least squares means = 0.3, 95% CI 2-sided [-0.1 to 0.7], Standard Error of Mean 0.23
Statistical Analysis 64: Comparison: Placebo vs Pregabalin 150 mg BID; Enjoyment of life: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.0002, ANCOVA; Difference in least squares means = -0.8, 95% CI 2-sided [-1.3 to -0.4], Standard Error of Mean 0.22
Statistical Analysis 65: Comparison: Placebo vs DS-5565 15 mg QD; Enjoyment of life: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.0271, ANCOVA; Difference in least squares means = -0.5, 95% CI 2-sided [-0.9 to -0.1], Standard Error of Mean 0.22
Statistical Analysis 66: Comparison: Placebo vs DS-5565 15 mg BID; Enjoyment of life: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.1123, ANCOVA; Difference in least squares means = -0.4, 95% CI 2-sided [-0.8 to 0.1], Standard Error of Mean 0.22
Statistical Analysis 67: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Enjoyment of life: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.1183, ANCOVA; Difference in least squares means = 0.3, 95% CI 2-sided [-0.1 to 0.8], Standard Error of Mean 0.22
Statistical Analysis 68: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Enjoyment of life: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.0299, ANCOVA; Difference in least squares means = 0.5, 95% CI 2-sided [0.0 to 0.9], Standard Error of Mean 0.22

12. Secondary Outcome: Proportion of Days a Rescue Medication Was Used in Participants Receiving DS-5565, Pregabalin, or Placebo
Description: Proportion of days with rescue medication intake during the double-blind treatment period equals number of days with rescue medication intake/(date of last study drug administration in the double-blind treatment period) - date of first study drug administration + 1).
Time Frame: Week 1 to Week 13 postdose
Population: Rescue medication usage was assessed using the modified intent-to-treat (mITT) analysis set.
Measure: Mean (Standard Deviation); unit: proportion of days
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
Number analyzed (Participants) | 315 | 312 | 315 | 313
proportion of days | 0.23 (0.32) | 0.21 (0.31) | 0.22 (0.32) | 0.21 (0.31)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin 150 mg BID; Test type: Superiority; p = 0.5578, ANCOVA; Difference in least squares means = -0.015, 95% CI 2-sided [-0.063 to 0.034], Standard Error of Mean 0.0249
Statistical Analysis 2: Comparison: Placebo vs DS-5565 15 mg QD; Test type: Superiority; p = 0.7034, ANCOVA; Difference in least squares means = -0.009, 95% CI 2-sided [-0.058 to 0.039], Standard Error of Mean 0.0248
Statistical Analysis 3: Comparison: Placebo vs DS-5565 15 mg BID; Test type: Superiority; p = 0.4143, ANCOVA; Difference in least squares means = -0.020, 95% CI 2-sided [-0.069 to 0.028], Standard Error of Mean 0.0249
Statistical Analysis 4: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg QD; Test type: Superiority; p = 0.8365, ANCOVA; Difference in least squares means = 0.005, 95% CI 2-sided [-0.044 to 0.054], Standard Error of Mean 0.0249
Statistical Analysis 5: Comparison: Pregabalin 150 mg BID vs DS-5565 15 mg BID; Test type: Superiority; p = 0.8189, ANCOVA; Difference in least squares means = -0.006, 95% CI 2-sided [-0.055 to 0.043], Standard Error of Mean 0.0249

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from baseline up to 4 weeks after the last study drug, up to 1 year 8 months.
Description: A TEAE is any adverse event that emerges on or after the first dosing of double blind study medication and during study treatment up to 4 weeks after the last dose of double blind study medication (having been absent prior to treatment) or worsens relative to the pre-double blind treatment state.
Arm/Group | Placebo | Pregabalin 150 mg BID | DS-5565 15 mg QD | DS-5565 15 mg BID
All-Cause Mortality (participants affected / at risk) | 0/315 | 0/312 | 1/315 | 0/313
Serious Adverse Events (participants affected / at risk) | 6/315 | 5/312 | 7/315 | 11/313
Other Adverse Events (participants affected / at risk) | 206/315 | 299/312 | 290/315 | 242/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=315) | Pregabalin 150 mg BID (N=312) | DS-5565 15 mg QD (N=315) | DS-5565 15 mg BID (N=313)
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 2
Mania (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Papilloedema (Eye disorders) | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=315) | Pregabalin 150 mg BID (N=312) | DS-5565 15 mg QD (N=315) | DS-5565 15 mg BID (N=313)
Weight increased (Investigations) | 9 | 39 | 17 | 33
Headache (Nervous system disorders) | 40 | 37 | 44 | 45
Dizziness (Nervous system disorders) | 23 | 47 | 44 | 41
Somnolence (Nervous system disorders) | 10 | 29 | 23 | 29
Vision blurred (Eye disorders) | 5 | 14 | 16 | 13
Drug withdrawal syndrome (General disorders) | 20 | 32 | 32 | 28
Fatigue (General disorders) | 9 | 11 | 17 | 11
Oedema peripheral (General disorders) | 4 | 10 | 9 | 16
Nausea (Gastrointestinal disorders) | 14 | 10 | 18 | 28
Diarrhoea (Gastrointestinal disorders) | 15 | 15 | 20 | 14
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 17 | 15 | 10 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 8 | 12 | 11
Nasopharyngitis (Infections and infestations) | 17 | 19 | 17 | 20
Urinary tract infection (Infections and infestations) | 6 | 13 | 11 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No